CLINICAL TRIAL: NCT05237622
Title: The FUNK-FLOW Study - Functional Residual Capacity During Different Levels of High-flow in Preterm Infants
Brief Title: Functional Residual Capacity During Different Levels of High-flow in Preterm Infants
Acronym: FunkFlow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FunkFlow
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Infant, Premature, Diseases; Respiratory Distress Syndrome
Keywords: Non-invasive respiratory support; HighFlow; continuous positive airway pressure; functional residual capacity
MeSH Terms: conditions — Infant, Premature, Diseases; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Flow (Other): Standard HighFlow therapy after weaning from continuous positive airway pressure therapy will be applied on different flow levels. Starting with a flow level of 8l/min, the flow-rates will be changed every 30 minutes subsequently from 8-6-4-2-4-6-8 l/min. Meanwhile, data lung volume changes will be measured using electrical impedance tomography.
  Interventions: Device: High Flow

INTERVENTIONS:
Device: High Flow — Standard HighFlow therapy after weaning from continuous positive airway pressure therapy will be applied on different flow levels. Starting with a flow level of 8l/min, the flow-rates will be changed every 30 minutes subsequently from 8-6-4-2-4-6-8 l/min. Meanwhile, data on lung volume changes will be measured using electrical impedance tomography.

SUMMARY:
Although there is a widespread use of HighFlow therapy around the world, there is still uncertainty about the most appropriate initial HighFlow level after nasal continuous positive airway pressure therapy. Higher levels might produce excessive and harmful intra-alveolar pressures exceeding those reached during nasal continuous positive airway pressure therapy. Low levels may not generate sufficient distending pressures, which may result in a loss of functional residual capacity and an increased risk of respiratory failure. Therefore, the aim of this study is to assess the effect of different HighFlow levels on the functional residual capacity and to compare these findings to the functional residual capacity during nasal continuous positive airway pressure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent by one or both parents or legal guardians as documented by signature
* 30 - 35 weeks postmenstrual age
* Respiratory support with nCPAP PEEP 5mbar and FiO2 < 0.30
* > 72 hours old

Exclusion Criteria:

* Inability of the parents to understand the study concept or procedures due to cognitive or linguistic reasons
* Congenital malformations adversely affecting lung aeration or pulmonary perfusion (e.g. congenital heart or lung defects)

Min Age: 73 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-19 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Change in global end-expiratory lung impedance (EELI) during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in global EELI over time using electrical impedance tomography (EIT)

SECONDARY OUTCOMES:
Change in mean respiratory rate (RR) during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in RR over time using electrical impedance tomography (EIT)
Change in regional end-expiratory lung impedance (EELI) during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in regional EELI over time using electrical impedance tomography (EIT)
Change in mean minute volume during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in mean minute volume over time using electrical impedance tomography (EIT), (AU/kg/min)
Change in mean ventilation distribution during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in mean ventilation distribution over time using electrical impedance tomography (EIT), (%, left/right and ventral/dorsal)
Change in mean silent spaces during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in mean silent spaces over time using electrical impedance tomography (EIT), (%, dependent, non-dependent lung)
Change in mean tidal volume during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in mean tidal volume over time using electrical impedance tomography (EIT), (AU/kg)
Change in number of apnoea that required stimulation during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in number of apnoea over time
Change in heart rate during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in heart rate over time
Change in oxygen saturation during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in oxygen saturation over time, SpO2, %
Change in fraction of inspired oxygen during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Change in fraction of inspired oxygen over time
Change in reaching 'failure criteria' to stop HighFlow therapy during the weaning procedure from nasal continuous positive airway pressure (nCPAP) to HighFlow (HF) | 230-minute recording period per patient, 30 minutes on each HF level
  Definition of failure criteria:
  * Respiratory rate > 100/min for at least 30 minutes during the intervention
  * Increase in FiO2 by ≥ 0.25 from baseline to maintain oxygen saturation level within physician-ordered parameters
  * > 2 apnoea requiring stimulation per 30-minute-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Newborn Research, Department of Neonatology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Collins CL, Holberton JR, Barfield C, Davis PG. A randomized controlled trial to compare heated humidified high-flow nasal cannulae with nasal continuous positive airway pressure postextubation in premature infants. J Pediatr. 2013 May;162(5):949-54.e1. doi: 10.1016/j.jpeds.2012.11.016. Epub 2012 Dec 20. PMID 23260098
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] van der Burg PS, Miedema M, de Jongh FH, Frerichs I, van Kaam AH. Cross-sectional changes in lung volume measured by electrical impedance tomography are representative for the whole lung in ventilated preterm infants. Crit Care Med. 2014 Jun;42(6):1524-30. doi: 10.1097/CCM.0000000000000230. PMID 24561568